CLINICAL TRIAL: NCT00015834
Title: A Phase I/II Trial of STI571 and High-Dose Cytarabine in Myeloid Blast Crisis of Chronic Myeloid Leukemia
Brief Title: STI571 Plus Cytarabine in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02374; UCLA-0011009; CDR0000068441 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Blastic Phase Chronic Myelogenous Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Cytarabine

ARMS (1):
- Treatment (imatinib mesylate, cytarabine) (Experimental): Patients who have not previously received imatinib mesylate receive oral imatinib mesylate daily on days 1-35. Patients who have previously received imatinib mesylate for at least 28 days receive oral imatinib mesylate on days 22-35. All patients receive cytarabine IV over 2 hours every 12 hours on days 29-32. Patients with more than 5% residual blasts in bone marrow on day 28 receive a second course in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Drug: cytarabine

INTERVENTIONS:
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside

SUMMARY:
Phase I/II trial to study the effectiveness of combining STI571 and chemotherapy in treating patients who have chronic myelogenous leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. STI571 may stop the growth of leukemia cells. Combining chemotherapy and STI571 may kill more cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of high-dose cytarabine when combined with imatinib mesylate in patients with blastic phase chronic myelogenous leukemia.

II. Determine the safety of this regimen in these patients. III. Determine the pharmacokinetics of this regimen in these patients. IV. Determine the frequency of hematologic and cytogenetic responses, duration of response, and survival of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of cytarabine.

Phase I: Patients who have not previously received imatinib mesylate receive oral imatinib mesylate daily on days 1-35. Patients who have previously received imatinib mesylate for at least 28 days receive oral imatinib mesylate on days 22-35. All patients receive cytarabine IV over 2 hours every 12 hours on days 29-32. Patients with more than 5% residual blasts in bone marrow on day 28 receive a second course in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of cytarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that which 2 of 6 patients experience dose-limiting toxicity.

Phase II: Additional patients are treated at the dose level preceding the MTD. Patients are followed monthly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic myelogenous leukemia in myeloid blast crisis

  * At least 30% blasts in bone marrow
* Philadelphia chromosome positive by cytogenetic analysis
* bcr/abl translocation by fluorescent in situ hybridization
* Ineligible for or refused allogeneic stem cell transplantation
* Not previously treated with imatinib mesylate OR currently receiving imatinib mesylate with stable disease on 2 bone marrow biopsies at least 2 weeks apart
* Performance status - ECOG 0-2
* See Disease Characteristics
* Bilirubin less than 3 times upper limit of normal (ULN)
* AST and ALT less than 3 times ULN
* Creatinine less than 2 times ULN
* No New York Heart Association class III or IV heart disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 2 weeks after study for female patients and at least 3 months after study for male patients
* See Disease Characteristics
* No prior allogeneic bone marrow or peripheral blood stem cell transplantation
* At least 48 hours since prior interferon alfa
* At least 24 hours since prior hydroxyurea
* At least 6 weeks since prior busulfan
* No other prior chemotherapy for blast crisis (except hydroxyurea)
* Concurrent hydroxyurea or anagrelide for severe leukocytosis or thrombocytosis allowed
* At least 4 weeks since prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2001-05; Primary Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Toxicity according to NCI/NIH Common Toxicity Criteria | Up to 2 years
  Described by duration, relatedness to treatment, and action taken.
Hematologic response | Up to 6 months
Bone marrow cytogenetic response | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Paquette, Principal Investigator — University of California at Los Angeles (UCLA )
Locations (1):
- University of California at Los Angeles (UCLA ), Los Angeles, California, United States